CLINICAL TRIAL: NCT00628615
Title: Non-Micturation Bladder Activity in Relation to Self-Consciousness During Filling Phase and Sensation Measurement During the Filling Phase
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Maastricht University, University hospital Maastricht
Other Study IDs: MEC 08-2-029
Record Dates: First submitted 2008-02-25; First posted 2008-03-05 (Estimated); Last update posted 2008-12-16 (Estimated); Status verified 2008-12

CONDITIONS: Lower Urinary Tract Symptoms; Overactive Bladder Syndrome
Keywords: Urodynamics; Overactive bladder syndrome; Lower urinary tract symptoms LUTS
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 2: male patients with lower urinary tract symptoms
- 1: Female patients with overactive bladder syndrome

SUMMARY:
Rationale:

The sensation of the need for urination (urge) is a complex and only partially understood mechanism. It is our hypothesis that this mechanism is disrupted in patients suffering from overactive bladder syndrome.

The Overactive Bladder syndrome (OAB) has been defined as a spectrum of symptoms in which incontinence may or may not overlap with urgency, frequency and nocturia. This syndrome is estimated to affect approximately 17% of the adult population in Europe and the United States. The symptoms of overactive bladder have many potential causes and contributing factors. One of these factors is an outlet obstruction of the bladder due to benign prostatic hyperplasia (BPH). Nowadays antimuscarinic drugs are used for treatment of the overactive bladder. Antimuscarinic agents have been proven to work slightly to moderately better than placebo's and are associated with side effects such as a dry mouth, blurred vision and constipation.

Many patients with lower urinary tract symptoms (LUTS) develop OAB. In this group of patients with LUTS and OAB, there is not always a clear obstruction found. So, at least in some patients, with LUTS, there must be another reason for OAB than obstruction.

The autonomous bladder activity has been introduced by, among others the Maastricht Urology research group. In animal models, the bladder is shown to have rhythmic low amplitude contractions (micro motions). It is hypothesized that this activity has a sensory function in the micturation regulation system which is mainly located in the bladder wall. These so called micromotions have never been demonstrated in the human bladder. The sensing function of the bladder and the micturation reflex remain mainly unclear. We hypothesise that there is a disregulation of the autonomous bladder activity (micro motions) in patients with OAB.

We want to explore and study the relationship between OAB, obstruction and the micro motions in order to gain a better understanding of the bladder (patho)physiology. reason for This on its turn, can help us in the quest for better treatment strategies for patients suffering from OAB.

Objective:

The study is divided in two distinct groups a male and female group:

The male group consist of patients with lower urinary tract symptoms (LUTS). The female group consist of patients with the overactive bladder syndrome OAB.

The primary objective of this pilot experiment is to describe via an observational study the relation between non-micturation bladder activity and sensation during the filling phase of the bladders in women. We want to explore if there is a relation between non-micturation bladder activity and the sensation of urgency during the filling phase.

Furthermore in men, we want to study the relationship between non-micturation bladder activity and the amount of obstruction.

We would also like to visualize the micro motions of the bladder in both men and women during filling phase and study the influence of (visual and cognitive) stimuli on bladder activity.

We want to explore if there is a relation between non-micturation bladder activity and the sensation of urgency during the filling phase in male patients with Lower urinary tract symptoms. In order to gain a better understanding in bladder (patho)physiology.

Study design: A pilot observational study to describe the non-micturation bladder activity and sensation measurement during filling phase.

Study population:

The study population consists of two groups. First a group of patients (female) who will undergo an ambulatory urodynamic investigation to investigate their bladder complaints. All patients will be older than 18 years.

The second group consists of male patients who will undergo a conventional urodynamic investigation in the normal work up for their lower urinary tract symptoms. All patients will be older than 18 years.

DETAILED DESCRIPTION:
Importance of the problem:

Incontinence, increased urge and increased frequency of micturition affect nearly 100 million people in the western world 1,2 (33 million in the US and 66 million in the European Union). These conditions are not life threatening but they seriously affect quality of life and ability to work. OAB is in some studies reported to have an incidence of up to 17 % in the western population with great consequences for the quality of life.

The lower urinary tract symptoms (LUTS) are more prevalent in the older population, where 40% over the age of 70 years are affected. Therefore, LUTS represent major problems to individuals, health professions and society. Importantly, as people are generally living longer, the numbers affected by LUTS are increasing.

Economic cost:

The total economic cost of this group of conditions is high. In 2002 the costs in the US were approximately $12.7 billion1 (estimated to be $17 billion and €22 billion/year in 2005). Approximately 25% of this expenditure is spent on treatment (drug therapy, clinical consultation and surgery). Of those who suffer only 28% have sought help and only half of those currently receive treatment. Less than 3% regain long lasting normal control. Therefore, these costs are an under-estimate and the problem is large.

Aetiology:

The primary clinical problem in the overactive bladder syndrome is an increased urge to pass urine, with or without incontinence. Remarkably, despite the prevalence and costs involved, the mechanisms underlying increased urge are not known. In order to simply describe the condition the term 'Over Active Bladder (OAB) Symptom Complex' has been introduced. In many cases, studied using conventional urodynamics, sensations of urge are correlated with rises in intra-vesical pressure, a condition classified as detrusor over activity (DO). In the remainder of patients, sensation is not accompanied by pressure changes and the condition can be described as bladder over activity (BO), previously described as sensory urgency. These differences in the relationship between sensation and bladder activity may be indicative of different clinical states. However, it is more likely that we don't yet understand the nature of the clinical condition.

Lower urinary tract symptoms are mostly caused by obstruction which is often caused by benign prostatic hypertrophia (BPH).

The study will be conducted among two distinct groups. a male and a female group.

The Female group:

In the female group the patients will be asked to describe their complaints while standard ambulatory urodynamic investigation takes place. Patients are asked to spend one hour of the six hours time which is the normal time for ambulatory urodynamics with us in the clinic.

During this time patients are asked to sit or stand up right and answer a few questions about their bladder sensations. Normally patients are free to go home and with this study these women are asked to spend the first hour in our clinic.

Patients will be asked to fill in a self-consciousness questionnaire in the period around the urodynamic measurement. They can do that before or after the measurement at home. This will take about 10 minutes.

Patients will also be asked to think of the answer to a few questions shown on a computer screen, during the urodynamic measurements. They will also be shown a few pictures, e.g. toilets or landscape pictures.

After obtaining informed consent, at the beginning of the normal procedure for a ambulatory urodynamic measurement the vesical catheter which is inserted in the patient for the purpose of the ambulatory urodynamic measurement will be connected to a more sensitive measuring device (PASAQ) with a 601 certification, designed by the IDDEE department of the Maastricht university and approved by the Maastricht university hospital technical department. (Mr. Frank Meeuwissen).

The bladder of the patient will be filled physiologically by the kidneys after drinking fluids, we will measure with a high sensibility, and try to study the small bladder contractions.

At intervals of 15 minutes the patient will be shown a computer screen on which 2 questions will be written. (e.g. Do you have a desire to void now?) the patient does not need to answer that question. We hypothesize that thinking of this question will trigger very small bladder contractions which allows the brain to , feel ' the bladder filling. The patient will also be shown a few pictures (e.g. a toilet and a landscape picture) in order to assess the effect of , and the difference between these visual stimuli on bladder contraction.

The male group:

In the study of male patients who are undergoing a standard stationary urodynamic measurement in the normal diagnostic work for their lower Urinary tract symptoms are asked to take part in the study.

This means that the measurement will take some 10 minutes more and that they are asked to fill in a questionnaire. There will be no extra catheter insertion or any invasive measurements added to the normal procedure of the conventional urodynamic measurements which they are undergoing for their symptoms.

Patients will be asked to fill in a self-consciousness questionnaire in the period around the urodynamic measurement. They can do that before or after the measurement at home. This will take about 10 minutes.

Patients will also be asked to think of the answer to a few questions shown on a computer screen, during the urodynamic measurements. They will also be shown a few pictures, e.g. toilets or landscape pictures.

We want to study the effect of such a visual or cognitive stimuli on the bladder contraction.

After obtaining informed consent, at the end of the normal procedure for a conventional urodynamic measurement the vesical catheter will remain in the patient for about ten minutes longer. This catheter is then connected to a more sensitive measuring device (PASAQ) with a 601 certification, designed by the IDDEE department of the Maastricht university and approved by the Maastricht university hospital technical department. (Mr. Frank Meeuwissen).

The bladder of the patient will be filled just like in a normal urodynamic measurement up to 3 different fillings, 100, 200 and 300 ml. At each of these filling amounts, the pomp will be stopped during 2 minutes and we will measure with a high sensibility, and try to study the small bladder contractions. At the 300 ml filling the patient will be shown a computer screen on which 2 questions will be written. (e.g. Do you have a desire to void now?) the patient does not need to answer that question. We hypothesise that thinking of this question will trigger very small bladder contractions which allows the brain to , feel ' the bladder filling. The patient will also be shown a few pictures (e.g. a toilet and a landscape picture) in order to assess the effect of , and the difference between these visual stimuli on bladder contraction.

Main study parameters/endpoints:

In the female group the main study parameters will be to characterize non-micturition activity during bladder filling in relation to visual and cognitive stimuli. This new high definition device will allow us to measure small an delicate changes in bladder pressure and allow us to relate this activity to bladder volume and sensation, to determine the nature of any change in this activity associated with OAB. The secondary study parameters are to identify possible mechanisms underlying OAB, to explore the possibility that therapeutically important drugs for OAB exert their action via inhibition of non-micturition activity

The main study parameters in the male group are to characterize non-micturition activity during bladder filling, to relate this activity to bladder volume and sensation, to determine the nature of any change in this activity associated with OAB and assess the relationship between the OAB symptoms with the amount of obstruction. The secondary study parameters are to identify possible mechanisms underlying OAB, to explore the possibility that therapeutically important drugs for OAB exert their action via inhibition of non-micturition activity.

Nature and extent of burden and risks associated with participation, benefit and group relatedness: Patients that participate in this study will not be exposed to serious adverse events and there will be no side effects. The investigation that they undergo for the normal workup of their complaints will take about ten minutes longer.

The patients will be asked to fill in an extra question list the so called self-consciousness questionnaire.

Patients will benefit of this study in directly, because it will be helpful in getting information on non-micturation activity and the relation with sensation. The results hopefully will lead to a better understanding of the normal and pathological bladder.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with lower urinary tract symptoms
* Female patients with overactive bladder syndrome

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male patients with lower urinary tract symptoms Female patients with overactive bladder syndrome
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
To characterise non-micturition activity during normal bladder filling | 2008-2009
To determine the nature of any change in this activity associated with OAB | 2008-2009
To relate this activity to bladder volume and sensation. | 2008-2009
To demonstrate the micromotions | 2008-2009
To study the link between OAB and micromotions in relation to bladder neck obstruction | 2008-2009

SECONDARY OUTCOMES:
To identify possible mechanisms underlying OAB | 2008-2009
To gain ideas for a better treatment for OAB | 2008-2009
To explore the possibility that therapeutically important drugs for OAB exert their action via inhibition of non-micturition activity | 2008-2009

CONTACTS AND LOCATIONS:
Overall Officials: Sajjad Rahnama'i, MD, Principal Investigator — Maastricht University Hospital; Gommert van koeveringe, MD, Study Director — Maastricht University Hospital
Locations (1):
- University Hospital Maastricht, Maastricht, Netherlands